CLINICAL TRIAL: NCT00656994
Title: A Phase III Safety Study to Evaluate the Long-term Effects of TAK-375 on Endocrine Function in Adult Subjects With Chronic Insomnia
Brief Title: Long-Term Efficacy of Ramelteon on Endocrine Function in Adult Subjects With Chronic Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-02-TL-375-032; U1111-1114-2594 (Registry Identifier: WHO)
Record Dates: First submitted 2008-03-12; First posted 2008-04-14 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia
Keywords: Sleep Disorder; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon 16 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 16 mg, tablets, orally, once nightly for up to 6 months.
  Other Names: Rozerem; TAK-375
  Arms: Ramelteon 16 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once nightly for up to 6 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the long-term effects of Ramelteon, once daily (QD), on endocrine function values.

DETAILED DESCRIPTION:
Insomnia is characterized by a complaint of either difficulties initiating and maintaining sleep or of nonrestorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had "ever had difficulty sleeping." Based on reports of "regular" or "frequent" sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is a melatonin-1 receptor agonist under global development by Takeda Chemical Industries, Ltd., Osaka, Japan, for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

This study has been designed to determine the long-term (6 month) effects of Ramelteon on endocrine function values. Study participation is anticipated to be about 7 months.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Has had primary insomnia as defined by the Diagnostic and Statistical Manual of Mental Disorders, Text Revision for at least 3 months and a history of daytime complaint(s) associated with disturbed sleep.
* Has a subjective sleep latency (sSL) greater than or equal to 45 minutes and a subjective total sleep time less than or equal to 6.5 hours for at least 3 nights out of one week.
* Habitual bedtime is between 8:30PM and 12:00AM.
* Habitual awakening time is between 5:00 AM and 10:00 AM.
* Male and female subjects must have serum prolactin, luteinizing hormone, follicle stimulating hormone, adrenocorticotropic hormone, thyroid stimulating hormone, triiodothyronine and thyroxine within normal range. Normal ranges for luteinizing hormone and follicle stimulating hormone for female subjects will be defined as the lowest value among the menstrual phases to the highest value among the menstrual phases.
* Body mass index between 18 and 34, inclusive.
* Male subjects must have serum testosterone values of greater than or equal to 150 ng per dL.
* Female subjects must have serum estradiol values within normal range.

Exclusion Criteria

* Known hypersensitivity to ramelteon or related compounds, including melatonin.
* Previously participated in a study involving ramelteon.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to Day 1, whichever is longer.
* Sleep schedule changes required by employment (eg, shift worker) within three months prior to Day 1, or has flown across greater than three time zones within seven days prior to screening.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to Day 1.
* Ever had a history of seizures, sleep apnea, chronic obstructive pulmonary disease, restless leg syndrome, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* History of psychiatric disorder (including anxiety or depression) within the past 12 months.
* History of drug addiction or drug abuse within the past 12 months.
* History of alcohol abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, Text Revision and/or regularly consumes 4 or more alcoholic drinks per day.
* Current significant neurological (including psychiatric and cognitive disorders), hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease, unless currently controlled and stable with protocol-allowed medication 30 days prior to Day 1.
* Uses tobacco products during nightly awakenings.
* Used melatonin, or other drugs or supplements known to affect sleep/wake function within 1week (or 5 half lives of the drug, whichever is longer) prior to Day 1.
* Used any central nervous system medication within 1 week (or 5 half lives of the drug, whichever is longer) prior to Day 1. These medications must not have been used to treat psychiatric disorders.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel including anti- hepatitis A virus (only immunoglobulin M is exclusionary), anti- hepatitis B surface (except in subjects who have received hepatitis B virus vaccination), hepatitis B surface antigen, anti-hepatitis B core (only immunoglobulin M is exclusionary), or anti-hepatitis C virus..
* Any significant endocrine pathology based on borderline laboratory results.
* Any additional condition(s) that in the Investigator's opinion would:

  * affect endocrine function (eg, hyperthyroidism, diabetes)
  * prohibit the subject from completing the study, or
  * not be in the best interest of the subject to participate in the study.
* Morning serum cortisol at the Screening visit of less than 7.0 μg per dl.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * anxiolytics
  * hypnotics
  * antidepressants
  * anticonvulsants
  * sedating H1 antihistamines
  * systemic steroids
  * respiratory stimulants (eg, theophylline) and decongestants
  * over-the-counter and prescription stimulants
  * over-the-counter and prescription diet aids
  * central nervous system active drugs
  * narcotic analgesics
  * beta blockers
  * St. John's Wort
  * kava-kava
  * gingko biloba
  * melatonin
  * other drugs or supplements known to affect sleep/wake function.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2003-01; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Total Serum Thyroxine. | Months 1, 2, 3, 4, 5, and 6 or Final Visit

SECONDARY OUTCOMES:
Change from baseline in free thyroxine. | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in thyroid stimulating hormone. | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in triiodothyronine. | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in total testosterone (men only). | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in free testosterone (men only). | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in estradiol (women only). | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in prolactin. | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in follicle stimulating hormone (women only). | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in luteinizing hormone (women only). | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in luteinizing hormone surge (women only) | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in adrenocorticotropic hormone. | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in cortisol (AM). | Months 1, 2, 3, 4, 5, and 6 or Final Visit
Change from baseline in adrenocorticotropic hormone stimulation test. | Month 6 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (29):
- United States (29):
  - Birmingham, Alabama
  - Jasper, Alabama
  - Mesa, Arizona
  - Peoria, Arizona
  - La Palma, California
  - Los Angeles, California
  - Riverside, California
  - San Diego, California
  - Denver, Colorado
  - Fort Lauderdale, Florida
  - West Palm Beach, Florida
  - Austell, Georgia
  - Roswell, Georgia
  - Des Moines, Iowa
  - Overland Park, Kansas
  - Prairie Village, Kansas
  - Florence, Kentucky
  - Wentzville, Missouri
  - Kenilworth, New Jersey
  - South Plainfield, New Jersey
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Ninety Six, South Carolina
  - Sioux Falls, South Dakota
  - Austin, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - Wichita Falls, Texas

REFERENCES:
- [Result] Richardson G, Wang-Weigand S. Effects of long-term exposure to ramelteon, a melatonin receptor agonist, on endocrine function in adults with chronic insomnia. Hum Psychopharmacol. 2009 Mar;24(2):103-11. doi: 10.1002/hup.993. PMID 19090503
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI